CLINICAL TRIAL: NCT01741467
Title: The Effect of Real Time Continuous Glucose Monitoring in Subjects With Pre-diabetes
Acronym: CGM PreDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Alicia L. Warnock, Director, Diabetes Institute, Walter Reed National Military Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 369196
Record Dates: First submitted 2012-07-19; First posted 2012-12-05 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pre-diabetes; Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RT-CGM (Experimental): Patients using the RT-CGM for the intervention portion of the study.
  Interventions: Behavioral: RT-CGM

INTERVENTIONS:
Behavioral: RT-CGM — Dexcom Seven+

SUMMARY:
This study will investigate whether real-time continuous glucose monitoring can be used as a tool for behavior change in people with pre-diabetes.

DETAILED DESCRIPTION:
The protocol is a prospective, non-blinded, randomized controlled study in persons with newly diagnosed pre-diabetes comparing the effects of real-time continuous glucose monitoring (RT-CGM) combined with diet and lifestyle education to those who have diet and lifestyle education alone. During a "wash-in" phase both groups will wear a masked CGM for 1 week at baseline and again after 12 weeks. Those randomized to the RT-CGM will wear it for 4 cycles of 2 week on/1 week off over the next 12 weeks. Both groups will follow-up with their primary care providers as clinically indicated over the next year with quarterly measurements of blood pressure, weight, and BMI. At the end of this period, they will wear a masked CGM for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Newly diagnosed with pre-diabetes (within the previous 6 months) with a FPG of > or = 110-125mg/dl or an A1c > or = 6% - 6.4%
* Able to independently measure and read finger stick blood glucose levels
* Willing to wear the CGM device for up to 12 weeks during the study period
* Willing to test blood sugar by fingerstick twice per day while wearing the CGM
* DEERS eligible

Exclusion Criteria:

* Using medication for pre-diabetes
* Women who are pregnant, lactating, planning to become pregnant, or without a safe contraceptive method; all female subjects will undergo pregnancy testing via a serum HcG with their initial blood testing.
* Subjects who are taking glucocorticoids, amphetamines, anabolic, or weight-reducing agents during the course of the study.
* Active Duty service members likely to be deployed during the 18-month study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Differences in blood glucose | baseline, 18 months
  Changes in A1c and fasting blood glucose over time and between the intervention and control groups.

SECONDARY OUTCOMES:
Impact of lifestyle changes | baseline, 18 months
  Evaluating the impact of lifestyle changes on levels of glycemic control in the control and experimental groups.
Changes in Glucose dynamics | baseline, 18 months
  Comparison of intervention and control group on standard measures of glucose dynamics.
Differences in blood pressure. | baseline, 18 months
  Objective comparison between the control and experimental group in changes in blood pressure.
Differences in lipids. | baseline, 18 months
  Objective comparison between the control group and the experimental group on changes in lipids.
Differences in weight | baseline, 18 months
  Objective comparison between the control group and the experimental group on changes in weight.
Changes in medication use | baseline, 18 months
  An objective comparison between the control and experimental group on changes in medication use.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vigersky, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Diabetes Prevention Program Research Group. The prevalence of retinopathy in impaired glucose tolerance and recent-onset diabetes in the Diabetes Prevention Program. Diabet Med. 2007 Feb;24(2):137-44. doi: 10.1111/j.1464-5491.2007.02043.x. PMID 17257275
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Yamaoka K, Tango T. Efficacy of lifestyle education to prevent type 2 diabetes: a meta-analysis of randomized controlled trials. Diabetes Care. 2005 Nov;28(11):2780-6. doi: 10.2337/diacare.28.11.2780. PMID 16249558
- [Background] Salpeter SR, Buckley NS, Kahn JA, Salpeter EE. Meta-analysis: metformin treatment in persons at risk for diabetes mellitus. Am J Med. 2008 Feb;121(2):149-157.e2. doi: 10.1016/j.amjmed.2007.09.016. PMID 18261504
- [Background] DeFronzo RA, Tripathy D, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Hodis HN, Kitabchi AE, Mack WJ, Mudaliar S, Ratner RE, Williams K, Stentz FB, Musi N, Reaven PD; ACT NOW Study. Pioglitazone for diabetes prevention in impaired glucose tolerance. N Engl J Med. 2011 Mar 24;364(12):1104-15. doi: 10.1056/NEJMoa1010949. PMID 21428766
- [Background] Chiasson JL. Acarbose for the prevention of diabetes, hypertension, and cardiovascular disease in subjects with impaired glucose tolerance: the Study to Prevent Non-Insulin-Dependent Diabetes Mellitus (STOP-NIDDM) Trial. Endocr Pract. 2006 Jan-Feb;12 Suppl 1:25-30. doi: 10.4158/EP.12.S1.25. PMID 16627376
- [Background] Van de Laar FA, Lucassen PL, Akkermans RP, Van de Lisdonk EH, De Grauw WJ. Alpha-glucosidase inhibitors for people with impaired glucose tolerance or impaired fasting blood glucose. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD005061. doi: 10.1002/14651858.CD005061.pub2. PMID 17054235
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Background] Battelino T, Phillip M, Bratina N, Nimri R, Oskarsson P, Bolinder J. Effect of continuous glucose monitoring on hypoglycemia in type 1 diabetes. Diabetes Care. 2011 Apr;34(4):795-800. doi: 10.2337/dc10-1989. Epub 2011 Feb 19. PMID 21335621
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Bode B, Beck RW, Xing D, Gilliam L, Hirsch I, Kollman C, Laffel L, Ruedy KJ, Tamborlane WV, Weinzimer S, Wolpert H. Sustained benefit of continuous glucose monitoring on A1C, glucose profiles, and hypoglycemia in adults with type 1 diabetes. Diabetes Care. 2009 Nov;32(11):2047-9. doi: 10.2337/dc09-0846. Epub 2009 Aug 12. PMID 19675193
- [Background] Vigersky RA, Fonda SJ, Chellappa M, Walker MS, Ehrhardt NM. Short- and long-term effects of real-time continuous glucose monitoring in patients with type 2 diabetes. Diabetes Care. 2012 Jan;35(1):32-8. doi: 10.2337/dc11-1438. Epub 2011 Nov 18. PMID 22100963
- [Background] Diabetes Prevention Program Research Group. The 10-year cost-effectiveness of lifestyle intervention or metformin for diabetes prevention: an intent-to-treat analysis of the DPP/DPPOS. Diabetes Care. 2012 Apr;35(4):723-30. doi: 10.2337/dc11-1468. PMID 22442395
- [Background] American Diabetes Association. Standards of medical care in diabetes--2011. Diabetes Care. 2011 Jan;34 Suppl 1(Suppl 1):S11-61. doi: 10.2337/dc11-S011. No abstract available. PMID 21193625